CLINICAL TRIAL: NCT00613444
Title: Photodynamic Therapy in the Treatment of Acne Vulgaris Using Non-Coherent Red Light (Derm 590)
Brief Title: Photodynamic Therapy in the Treatment of Acne
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never started due to logistical issues.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey S. Orringer, Professor of Dermatology, Medical School, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Derm 590; HUM00016677
Record Dates: First submitted 2008-01-30; First posted 2008-02-13 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Acne Vulgaris
Keywords: Acne; laser
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- LumaCare LC-122M non-coherent light source (Experimental): Split Face Comparison. One half of subject's face will receive topical photosensitizer applications followed by LumaCare LC-122M non-coherent light source illumination. Subjects will receive a series of up to 6 treatment sessions with a treatment interval of from approximately 1 to 4 weeks. In all cases, light treatment parameters will be within the guidelines normally used clinically for red-light non-coherrent light sources, and thus fluences used will not exceed 75 J/cm2.
  The other half of the face will not receive any treatment and will serve as internal control.
  Interventions: Device: LumaCare LC-122M non-coherent light source

INTERVENTIONS:
Device: LumaCare LC-122M non-coherent light source — Subjects will receive a series of up to 6 treatment sessions with a treatment interval of from approximately 1 to 4 weeks. In all cases, light treatment parameters will be within the guidelines normally used clinically for red-light non-coherrent light sources, and thus fluences used will not exceed 75 J/cm2.

SUMMARY:
The purpose of this research project is to study the effect of non-ablative (non-cutting) laser therapy, a technique that uses laser energy to try to improve the appearance of the skin. This type of laser treatment creates changes in a layer of the skin called the dermis without causing an open wound in the skin. The use of non-ablative laser therapy, together with application of a photo-sensitizer (substance that makes the skin more sensitive to light), may improve the appearance of acne. The idea behind the photo-sensitizer is that it is supposed to make the laser more effective than using just the laser alone. It is not yet clear how much improvement can be seen with these treatments or exactly how the skin's response causes these improvements. In this study, we are interested in learning how well such a laser works to improve the symptoms of acne, as well as how much the photo-sensitizer actually enhances the efficacy of the laser.

The photo-sensitizing agent (Levulan Kerastick) and the non-ablative laser (LumaCare LC-122M non-coherent (multiple wavelengths) light source from LumaCare® Medical Products) are both FDA-approved. The Levulan Kerastick is approved for the treatment of another skin disease, not acne.

DETAILED DESCRIPTION:
Background

Acne vulgaris remains among the most common cutaneous disorders, impacting the vast majority of people at some point during their lives. It is associated with significant psychosocial morbidity, and there remains the need for efficacious and low risk therapeutic options.

The FDA has approved various lasers and light sources for the treatment of acne. However, few randomized, controlled clinical trials have been performed of these devices. In addition, the use of topical photosensitizers preceding laser or light-therapy for acne has also been examined in a preliminary way with some initial evidence of efficacy. However, these trials have been small with modest numbers of subjects, many focus on back acne, and treatment protocols vary widely and are often poorly controlled. Photodynamic therapy for facial acne is being performed by physicians across the country but little objective data regarding this practice is available.

We have recently conducted a trial of a 1 hour application of a common photosensitizer approved by the FDA for acne phototherapy (Levulan, DUSA pharmaceutical) using a pulsed dye laser therapy (V-Beam laser, Candela Corp., Wayland, MA, 595 nm wavelength) as the activating light source (IRB protocol 2005-0117). Interim results from our study indicate this therapy is effective in a minority of patients. Accumulating published reports data suggests the limited effectiveness of this protocol may be due to inadequate skin penetration of the photosensitizing agent and due to the need for an activating light source with a longer wavelength of light to allow deeper penetration into the skin. We wish to incorporate these findings to design a protocol that should be more effective for treatment of facial acne.

Objectives

We propose to evaluate the efficacy and confirm the safety of an FDA-approved non-coherent light source (LumaCare LC-122M non-coherent light source with LUM-I, fiber optic probe, 610 nm-660 nm output range, LumaCare Medical Products, Newport Beach, Ca) used in conjunction with a topical photosensitizer (Levulan, DUSA pharmaceutical) in the treatment of acne vulgaris. Because one proposed mechanism of action for such treatments includes altered sebaceous gland activity, we also seek to examine the effects of this treatment on cutaneous sebum production.

ELIGIBILITY:
Inclusion Criteria:

1. Age 15 years or older of either gender and of any racial/ethnic group.
2. Presence of clinically-evident facial acne.
3. Subjects must be in generally good health.
4. Subjects must be able and willing to comply with the requirements of the protocol.
5. Subjects must have Fitzpatrick skin type I, II or III.
6. You must live within a reasonable driving distance of Ann Arbor, Michigan, and/or be able to attend all of the scheduled appointments during the study.

Exclusion Criteria:

1. Oral retinoid use within six months of entry into the study.
2. Systemic acne therapies (oral antibiotics) within 4 weeks of entry into the study.
3. Topical acne therapies (retinoids, antibiotics) within 2 weeks of entry into the study.
4. Microdermabrasion or superficial chemical peels at the sites to be treated within 2 months of entry into the study.
5. Subjects with a history of dermabrasion or laser resurfacing at the sites to be treated.
6. Use of topical lipid absorbing substances (Clinac AC) within 2 weeks of entry into the study.
7. Non-compliant subjects.
8. Subjects with a significant medical history or concurrent illness/condition which the investigator(s) feel is not safe for study participation.
9. Subjects using alcohol-based topical solutions or "exfoliating" agents within 2 weeks of entry into the study.
10. Subjects with a history of very frequent herpes simplex infections of the face or with clinical evidence of active herpes simplex infections.
11. History of keloid scar formation for subjects undergoing biopsies.
12. Pregnant or nursing females.
13. Subjects with known allergy or hypersensitivity to topical photosensitizing agents.
14. Subjects with known photosensitivity disorders felt by the investigators to preclude safe inclusion in the study.
15. Subjects with Fitzpatrick skin type IV or greater.
16. Subjects who have a history of significant post-inflammatory hyperpigmentation at the sites of acne lesions.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2008-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Subtypes of acne lesions including papules, pustules, cysts, open comedones, and closed comedones. In addition to lesion counts, overall acne severity will be graded by the investigator using the Leeds acne severity scale. | Baseline and follow-up evaluations

SECONDARY OUTCOMES:
Sebum production | Baseline and follow-up evaluations
Photographs | Baseline and follow-up evaluations

CONTACTS AND LOCATIONS:
Overall Officials: John J Voorhees, MD, Study Chair — University of Michigan